CLINICAL TRIAL: NCT00337285
Title: A Long-Term, Open-Label, and Single-Arm Study of NRP104 30 mg, 50 mg, or 70 mg Per Day in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: An Open-label Study of NRP104 in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: New River Pharmaceuticals (Industry)
Collaborators: Shire (Industry)
Responsible Party: Timothy Whitaker, M.D., Shire Pharmaceutical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NRP104.304
Record Dates: First submitted 2006-06-09; First posted 2006-06-15 (Estimated); Results first posted 2009-07-17 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Attention Deficit Hyperactivity Disorder; Attention Deficit Disorders With Hyperactivity; Attention Deficit Hyperactivity Disorders
Keywords: Attention Deficit Hyperactivity Disorder; Attention Deficit Disorders with Hyperactivity; Attention Deficit Hyperactivity Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Vyvanse (lisdexamfetamine dimesylate), NRP104

INTERVENTIONS:
Drug: Vyvanse (lisdexamfetamine dimesylate), NRP104 — NRP104 capsule once-a-day orally beginning at 30mg/day and titrated by 20 mg per day at weekly intervals up to a maximum daily dose of 70 mg

SUMMARY:
The purpose of this study is to assess the long-term safety and efficacy of three NRP104 doses of 30 mg, 50 mg, or 70 mg, administered at the same time daily, in the treatment of adults with ADHD.

DETAILED DESCRIPTION:
This is a multi-center, open-label, and single-arm study to assess the safety of three NRP104 doses (30 mg, 50 mg, or 70 mg per day) for up to one (1) year in the treatment of adults with ADHD. Subjects who were randomized and met all inclusion/exclusion criteria in Protocol NRP104.303 are eligible for participation in this protocol. The study will consist of three periods: a screening/baseline period, a 4-week dose titration, and a long-term maintenance of up to 11 months. There are three possibilities for subjects that rollover from the NRP104.303 protocol. They are:

Subjects that rollover at the final visit of the NRP104.303 study (on the same day):

The screening and baseline procedures from this open label study will coincide with the final study visit of Protocol NRP104.303. Subject data from final study visit will be transferred and utilized for the open label study. On this same day, the subject will be consented for NRP104.304, inclusion/exclusion criteria will be assessed, the subject will be enrolled, and study medication will be dispensed.

Subjects that rollover not on the same day but within seven days of the NRP104.303 study:

If the subject returns to enroll into the NRP104.304 study within seven days of the final NRP104.303 study visit and has not taken any excluded medications for which a washout is required, the final study visit procedures and data from the NRP104.303 study will be transferred and utilized for the screening and baseline visit procedures of this study, where applicable. When the subject returns to the site, they will be consented, inclusion and exclusion criteria will be assessed, the subject will be enrolled, and study medication will be dispensed.

Subjects will require a full screening visit if more than 7 days have elapsed since they completed the NRP104.303 study:

After screening results have been received by the site, the site personnel will contact the subject via telephone to inform them of continued study eligibility. During this call the subject will be instructed to stop all medications for the treatment of ADHD, if any. This call starts the washout of all psychoactive medications, which should last 7 (±2) days. During the Washout Phone Contact, the visit dates for the Baseline visit (Visit 01) and Visits 02 through 05 should be scheduled at 7-day intervals as calculated from Baseline. After the washout is complete, subjects will return to the clinic for the baseline visit (Visit 01) to have the baseline procedures performed and to receive study medication.

Dose Titration

All subjects will initiate treatment at NRP104 30 mg for the 1st week. At the subsequent 4 weekly visits (Visits 02, 03, 04, and 05), the subject's daily dose of NRP104 may be increased or decreased by 20 mg at weekly intervals to achieve the optimal efficacy and tolerability, if deemed appropriate by the Investigator. In this study, the maximum daily dose of NRP104 that can be received by the subject is 70 mg, and the minimum daily dose of NRP104 the subject must take to continue the treatment is 30 mg.

Monthly Maintenance

At the end of the initial 4-week dose titration (Visit 05), subjects will enter the long-term maintenance of up to 11 months. Monthly visits, starting with Visit 06, will have a window of ±4 days. All visits will be scheduled relative to the Baseline Visit date. The last scheduled visit of the protocol is Visit 16 at Month 12. During the long-term maintenance, the subject's dose may be increased or decreased by 20 mg at any visit, if deemed appropriate by the Investigator, to maintain optimal treatment in terms of efficacy and tolerability. All reasons for dose changes should be well documented by the investigator during the maintenance period. Subjects who cannot maintain the minimum daily dose of NRP 30 mg due to intolerance will be withdrawn from the study.

Safety and Efficacy Assessments

ADHD Rating Scale (ADHD-RS) performed using adult prompts and Clinical Global Impression (CGI) will be assessed by the Investigator. The Pittsburgh Sleep Quality Index (PSQI) will be assessed once every three months following baseline.

Adverse events and concomitant medications will be recorded at each visit starting from the baseline visit. Vital signs will be measured at each visit from the screening visit. Physical exam and clinical laboratory tests (including pregnancy tests) will be assessed at Screening, Visit 10 and the final visit. Weight will be measured at the screening visit, baseline visit, and every month thereafter. Height will be measured at the screening visit and final visit. ECG parameters will be assessed at the screening visit, baseline visit, and every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18-55 years of age, inclusive, at the time of consent of the NRP104.303 study.
* Subject must have been randomized and must have met all inclusion/exclusion criteria in the NRP104.303 study.
* Subject must be male or non-pregnant female. Females of childbearing potential (FOCP) must comply with contraceptive restrictions noted in the protocol.
* Subject must have a satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, PE, clinical and laboratory evaluation.
* In the opinion of the investigator, the subject understands and is able, willing, and likely to fully comply with the study procedures and restrictions.
* Subject must have given written, personally signed and dated informed consent to participate in the study in accordance with the International Conference on Harmonization (ICH) Good Clinical Practice (GCP) Guidelines and applicable regulations before completing any study specific procedures.
* Subject experienced no adverse events in a previous study of NRP104 or elsewhere that would preclude continued exposure to NRP104.

Exclusion Criteria:

* Subject has any concurrent chronic or acute illness or unstable medical condition that could confound the results of safety assessments, increase risk to the subject or lead to difficulty complying with the protocol. Subjects who have a history of mental retardation or a severe learning disability are excluded.
* Subject has a known cardiac structural abnormality or any other condition that may affect cardiac performance.
* Subject has any clinically significant ECG or laboratory abnormality known to the investigator prior to dispensation of study medication.
* Subject has a resting sitting systolic blood pressure or diastolic blood pressure deemed clinically significant by the investigator.
* Subject has used any prohibited prescription medication except for medications used to treat ADHD within 30 days of screening visit. Hormonal contraceptives are acceptable.
* Subject has a positive urine drug result at Screening (with the exception of subject's current stimulant therapy, if any).
* Subject has taken an investigational drug or taken part in a clinical trial within 30 days prior to Screening (except for participating in an NRP104 study).
* The female subject is pregnant or lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 349 (Actual)
Dates: Start 2006-07; Primary Completion 2007-11 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Biederman, M.D., Principal Investigator — Massachusetts General Hospital
Locations (45):
- United States (45):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Valley Clinical Research, Inc., El Centro, California
  - University of California, Irvine Child Development Center, Irvine, California
  - Bay Area Research Institute, Lafayette, California
  - Peninsula Research Associates, Rolling Hills Estate, California
  - University of California, San Francisco, Dept. of Psychiatry, San Francisco, California
  - Encompass Clinical Research, Spring Valley, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Psychiatric Medicine Center, New London, Connecticut
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Miami Research Associates, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Meridien Research, Tampa, Florida
  - Janus Center for Psychiatric Research LLC, West Palm Beach, Florida
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Carman Research, Smyrna, Georgia
  - Psychiatric Associates, Overland Park, Kansas
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Johns Hopkins at Green Spring Station, Lutherville, Maryland
  - Marc Hertzman, MD, Rockville, Maryland
  - Masschusetts General Hospital, Cambridge, Massachusetts
  - Summit Research Network (Michigan) Inc., Flint, Michigan
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - St Charles Psychiatric Associates-Midwest Research, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Las Vegas, Nevada
  - CNS Research Institute (CRI), Clementon, New Jersey
  - VA New York Harbor Healthcare System, New York, New York
  - Duke University ADHD Program, Durham, North Carolina
  - Richard Weisler and Associates, Raleigh, North Carolina
  - The Ohio State University, Columbus, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - CNS Research Institute, P.C., Philadelphia, Pennsylvania
  - FutureSearch Trials, Austin, Texas
  - Claghorn-Lesem Research Clinic, Bellaire, Texas
  - Bayou City Research, Houston, Texas
  - Red Oak Psychiatry Associates, P.A., Houston, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - John M. Turnbow, MD, PA, Lubbock, Texas
  - The Clinical Study Center, Burlington, Vermont
  - Neuropsychiatric Associates, Woodstock, Vermont
  - Psychiatric Alliance of the Blue Ridge Clinical Research, Charlottesville, Virginia
  - NeuroScience, Inc., Herndon, Virginia
  - Brighton Research Group, Virginia Beach, Virginia
  - Summit Research Network LLC (Seattle), Seattle, Washington

REFERENCES:
- [Result] Ginsberg L, Katic A, Adeyi B, Dirks B, Babcock T, Lasser R, Scheckner B, Adler LA. Long-term treatment outcomes with lisdexamfetamine dimesylate for adults with attention-deficit/hyperactivity disorder stratified by baseline severity. Curr Med Res Opin. 2011 Jun;27(6):1097-107. doi: 10.1185/03007995.2011.567256. Epub 2011 Mar 28. PMID 21438796
- [Result] Mattingly G, Weisler R, Dirks B, Babcock T, Adeyi B, Scheckner B, Lasser R. Attention deficit hyperactivity disorder subtypes and symptom response in adults treated with lisdexamfetamine dimesylate. Innov Clin Neurosci. 2012 May;9(5-6):22-30. PMID 22808446
- See also: (FDA Recall Information) — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects received a 30, 50, or 70 mg once daily dose of Vyvanse for up to 1 year.
Groups:
- Vyvanse: Subjects received a 30, 50, or 70 mg once daily dose of Vyvanse (Lisdexamfetamine dimesylate) for up to 1 year.
Period: Overall Study
Arm/Group | Vyvanse
Started | 349
Completed | 191
Not Completed | 158
Not completed — Withdrawal by Subject | 42
Not completed — Lost to Follow-up | 41
Not completed — Adverse Event | 28
Not completed — Protocol Violation | 27
Not completed — Lack of Efficacy | 11
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Lack of protocol compliance | 7

BASELINE CHARACTERISTICS:
Arm/Group | Vyvanse
Number analyzed (Participants) | 349
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 349
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.8 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159
  Male | 190
Region of Enrollment [Number; unit: participants]
  United States | 349

OUTCOME MEASURES:

1. Primary Outcome: Change in ADHD-RS-IV Total Score From Baseline at Up to One Year
Description: Change in the Attention Deficit Hyperactivity Disorder Rating Scale-fourth edition (ADHD-RS-IV) total score from baseline. The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: up to one year
Population: Intent-to-treat (ITT). Defined as all subjects who were treated and had both the baseline and at least one post-baseline primary efficacy measurement (i.e., ADHD-RS-IV total score)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vyvanse
Number analyzed (Participants) | 345
Units on a scale | -24.8 (11.7)
Statistical Analysis 1: Comparison: Vyvanse; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Improvement on CGI-I
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement includes 1 and 2 on the scale.
Time Frame: Up to 1 year
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Vyvanse
Number analyzed (Participants) | 345
Participants | 290

3. Secondary Outcome: Change in PSQI Total Score From Baseline at Up to One Year
Description: Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire consisting of 18 items which generates seven component scores on a scale from 0 (better sleep) to 3 (worse sleep) resulting in a global score of 0-21, where a higher number reflects worse sleep quality.
Time Frame: up to 1 year
Population: Safety population (Defined as all subjects who were enrolled and who received at least one dose of the investigational product.)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Vyvanse
Number analyzed (Participants) | 349
Units on a scale | -1.3 (2.8)
Statistical Analysis 1: Comparison: Vyvanse; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Vyvanse
Serious Adverse Events (participants affected / at risk) | 8
Other Adverse Events (participants affected / at risk) | 306
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Vyvanse
Chest pain (Musculoskeletal and connective tissue disorders) | 1/349
Anal fissure (Gastrointestinal disorders) | 1/349
Cocaine and alcohol toxicity (Social circumstances) | 1/349
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/349
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1/349
Foot fracture (Injury, poisoning and procedural complications) | 1/349
Cholecystitis acute (Hepatobiliary disorders) | 1/349
Arthritis bacterial (Infections and infestations) | 1/349
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Vyvanse
Upper respiratory tract infection (Infections and infestations) | 76/349
Insomnia (Psychiatric disorders) | 68/349
Headache (Nervous system disorders) | 60/349
Dry mouth (Gastrointestinal disorders) | 58/349
Decreased appetite (Metabolism and nutrition disorders) | 50/349
Irritability (General disorders) | 39/349
Anxiety (Psychiatric disorders) | 29/349
Nasopharyngitis (Infections and infestations) | 26/349
Sinusitis (Infections and infestations) | 23/349
Weight decreased (Investigations) | 21/349
Back pain (Musculoskeletal and connective tissue disorders) | 19/349
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18/349

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.